CLINICAL TRIAL: NCT03141151
Title: Competency-based Approaches to Community Health
Acronym: COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Bill Heerman, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 170420
Record Dates: First submitted 2017-05-01; First posted 2017-05-04 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and data collectors will be blinded to randomization status. Because this is a behavioral intervention, the participants and interventionists will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COACH: Healthy Bodies (Experimental): This will be a staged intensity behavioral intervention. The intensive phase will last 15 weeks and consist of weekly, 90 minute, skills-building sessions. The content will focus on diet, physical activity, sleep, media use, and parenting. Behavior change techniques will include goal-setting, self-monitoring, and problem solving. Following the intensive phase, participants will enter a maintenance phase, consisting of monthly phone calls from a health coach for 3 months.
  Interventions: Behavioral: COACH: Healthy Bodies
- COACH: Strong minds (Active Comparator): This will be a school-readiness intervention for the 3-5 year old children involved, which will meet twice a month for 3 months. Group sessions will focus on building social support around literacy skills for parents and children, as well as school advocacy.
  Interventions: Behavioral: COACH: Strong Minds

INTERVENTIONS:
Behavioral: COACH: Healthy Bodies — Staged intensity behavioral intervention focusing on healthy lifestyles in the context of family.
  Arms: COACH: Healthy Bodies
Behavioral: COACH: Strong Minds — School Readiness Intervention focusing on literacy and parent skills
  Arms: COACH: Strong minds

SUMMARY:
This study is a family-centered, community-based intervention to prevent and treat childhood obesity among 3-5 year old children from undeserved communities. Half of participants will receive a healthy lifestyle intervention and half of participants will receive a school-readiness intervention.

DETAILED DESCRIPTION:
The complex multi-level determinants of childhood obesity necessitate a personalized approach. One of the main challenges to effective behavior change interventions is the complexity of the systems in which these behaviors are situated. Namely, health behaviors are the result of the confluence of macro-level influences (e.g., the built environment, family, etc.) and micro-level influences (e.g., stress). Furthermore, it is imperative that attempts to support healthy childhood growth consider the foundational contribution of a person's culture to their health behaviors, especially as children from traditionally underserved minorities are often hardest hit by obesity.

This program will test a 15 week behavioral intervention followed by 3 months of coaching calls that uses principles from the learning sciences and health behavior change to help shape healthy behaviors in the context of family. The follow-up of the study will last 1 year. The content of the intervention will focus on health behavior change, including teaching goal-setting and self monitoring skills, as well as parenting strategies.

The primary outcome of interest will be early childhood BMI trajectory over 1 year. Additional measures will include survey data to measure parent and child health behaviors (e.g., diet, physical activity, sleep, media use) that are associated with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Three-to-five year old child
2. Spanish or English-speaking
3. Child's BMI ≥ 50%
4. Parental commitment to participate in a year long study
5. Consistent phone access
6. Parent age ≥ 18 years
7. Child completion of baseline data collection on height, weight, and waist circumference and all willing survey items completed by the parent
8. Parents and children must be healthy (parents with controlled medical conditions will also be eligible).
9. Dyad must be considered underserved which will be indicated by the parents self-reporting if they or someone in their household participate in one of these programs or services: TennCare, CoverKids, WIC, Food Stamps (SNAP), Free and Reduced Price School Lunch and Breakfast, Families First (TANF), and/or subsidized housing

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Heerman, MD MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heerman WJ, Teeters L, Sommer EC, Burgess LE, Escarfuller J, Van Wyk C, Barkin SL, Duhon AA, Cole J, Samuels LR, Singer-Gabella M. Competency-Based Approaches to Community Health: A Randomized Controlled Trial to Reduce Childhood Obesity among Latino Preschool-Aged Children. Child Obes. 2019 Dec;15(8):519-531. doi: 10.1089/chi.2019.0064. Epub 2019 Aug 5. PMID 31381365
- [Derived] Adams LE, Sommer EC, Truesdale KP, Barkin SL, Heerman WJ. Validation of a new scoring approach of a child dietary questionnaire for use in early childhood among low-income, Latino populations. BMC Nutr. 2022 Oct 31;8(1):125. doi: 10.1186/s40795-022-00618-4. PMID 36316788

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds
Started | 59 | 58
Completed | 53 | 54
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 58 | 117
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (0.8) | 4.2 (0.8) | 4.2 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 27 | 27 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 59 | 58 | 117
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 117

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Body Mass Index
Description: child BMI trajectory across 12 months; BMI differences over time are estimates from the longitudinal mixed-effects regression model
Time Frame: Baseline, 4 months, 7 months, 1 year
Population: Number analyzed differs across each time point as it relates to retention
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds
Number analyzed (Participants) | 59 | 58
kg/m^2
  Baseline | 18.1 (2.2) | 18.1 (3.0)
  4 months: number analyzed (Participants) | 56 | 56
  4 months | 18.1 (2.5) | 18.2 (3.4)
  7 months: number analyzed (Participants) | 52 | 55
  7 months | 18.0 (2.5) | 18.4 (3.3)
  12 months: number analyzed (Participants) | 52 | 54
  12 months | 18.5 (2.7) | 18.7 (3.7)

2. Secondary Outcome: Child Diet: Soda
Description: Parent-reported survey data; Child diet: Soda was measured by a single survey item used in the Feeding Infants and Toddlers Study with higher values representing higher frequency of consumption per day. (citation: Ziegler P, Briefel R, Clusen N, et al. Feeding Infants and Toddlers Study (FITS): Development of the FITS survey in comparison to other dietary survey methods. J Am Diet Assoc 2006;106:S12-S27.)
Time Frame: 4 months
Population: Secondary analysis was based on participants with complete data on the Child Diet: Soda measure at baseline and 4 month follow-up timepoints. Note: number of participants analyzed differs slightly from the primary analysis of the primary outcome which was Child BMI.
Measure: Mean (Standard Deviation); unit: Sodas/day
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds
Number analyzed (Participants) | 56 | 55
Sodas/day | 0.17 (0.27) | 0.19 (0.31)

3. Secondary Outcome: Child Physical Activity
Description: Parent-reported survey data
Time Frame: 4 months
Population: Secondary analysis was based on participants with complete data on the child active days per week measure at baseline and 4 month follow-up timepoints. Note: number of participants analyzed differs slightly from the primary analysis of the primary outcome which was Child BMI.
Measure: Mean (Standard Deviation); unit: Child active days per week
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds
Number analyzed (Participants) | 55 | 55
Child active days per week | 2.00 (2.60) | 1.62 (2.63)

4. Secondary Outcome: Parent BMI
Time Frame: 4 months
Population: Secondary analysis was based on participants with complete data on the Adult BMI measure at baseline and 4 month follow-up timepoints. Note: number of participants analyzed differs slightly from the primary analysis of the primary outcome which was Child BMI.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds
Number analyzed (Participants) | 50 | 49
kg/m^2 | 30.44 (5.86) | 31.57 (6.72)

5. Secondary Outcome: Parent Diet Practices
Description: Self-reported survey data; Parent diet practices were measured by using a summed score of a 4-item questionnaire of eating behaviors, including overeating, unplanned eating, making poor food choices, and emotional eating. Higher scores represent more unhealthy parent dieting practices. Items ranged on a scale from 0-5 and were summed to create the scale which ranged from 0-20.
Time Frame: 4 months
Population: Secondary analysis was based on participants with complete data on the Parent Diet Practices measure at baseline and 4 month follow-up timepoints. Note: number of participants analyzed differs slightly from the primary analysis of the primary outcome which was Child BMI.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds
Number analyzed (Participants) | 55 | 54
score on a scale | 5.04 (4.09) | 5.22 (4.02)

6. Secondary Outcome: Parenting Practices: Engagement
Description: Self-reported survey data; Parenting practices around child physical activity were measured by the Preschooler Physical Activity Parenting Practices (PPAPP) scale which has an engagement subscale. Parenting practices: Engagement was a 15 item subscale of the PPAPP survey with higher scores representing higher parent engagement practices. Items ranged on a scale from 1-5 and were summed to create the subscale which ranged from 15-75.
Time Frame: 4 months
Population: Secondary analysis was based on participants with complete data on the Parent Practices: Engagement measure at baseline and 4 month follow-up timepoints. Note: number of participants analyzed differs slightly from the primary analysis of the primary outcome which was Child BMI.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds
Number analyzed (Participants) | 56 | 54
score on a scale | 53.79 (12.66) | 49.52 (13.06)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected throughout the study. We specifically asked about adverse events and serious adverse events at each follow-up time point (4 months, 7 months, 1 year), but always completed follow-up and documentation for any event in between data collection time points.
Arm/Group | COACH: Healthy Bodies | COACH: Strong Minds
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58
Other Adverse Events (participants affected / at risk) | 0/59 | 0/58

LIMITATIONS AND CAVEATS:
The study was conducted among Latino families; findings should not be generalized to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT03141151/Prot_SAP_000.pdf